CLINICAL TRIAL: NCT00243711
Title: A Multi-Center Randomized Study to Evaluate the Efficacy and Safety of an Investigational Lubricant Eye Drop
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG9689-001
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium; Glycerol

INTERVENTIONS:
Drug: Carboxymethylcellulose sodium and Glycerin

SUMMARY:
The efficacy, safety and acceptability of an investigational lubricant eye drop in subjects with dry eye will be evaluated in comparison with currently-available lubricant eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Mild, Moderate, or Severe Dry Eye Symptoms and current eye drop use;
* Reduced tear stability or tear production

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2005-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Dry Eye Symptoms

SECONDARY OUTCOMES:
Ocular surface damage, tear stability, tear production

CONTACTS AND LOCATIONS:
Overall Officials: Mark Curtis, O.D., Principal Investigator — InSight Eyecare
Locations (1):
- Warrensburg, Missouri, United States